CLINICAL TRIAL: NCT01179646
Title: A Pharmacokinetic Study to Determine the Bioequivalence of a Test 40 mg Pantoprazole Delayed-Release Tablet, Compared to a Marketed 40 mg Pantoprazole Delayed-Release Tablet (Protonix, Wyeth Pharmaceuticals) When Administered to Healthy Adult Subjects in the Fasted State
Brief Title: Bioequivalence Study of Pantoprazole 40 mg DR Tablets and Protonix 40 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kremers Urban Development Company (Industry)
Responsible Party: Alan S. Marion, MD, PhD, MDS Pharma Services (US) Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP796
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalency
MeSH Terms: interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protonix (Active Comparator): Protonix 40 mg DR Tablet
  Interventions: Drug: Pantoprazole 40 mg DR Tablet vs. Protonix 40 mg DR Tablet
- Pantoprazole (Experimental): Pantoprazole 40 mg DR Tablet
  Interventions: Drug: Pantoprazole 40 mg DR Tablet vs. Protonix 40 mg DR Tablet

INTERVENTIONS:
Drug: Pantoprazole 40 mg DR Tablet vs. Protonix 40 mg DR Tablet — Single dose crossover BE study
  Other Names: Protonix 40 mg DR Tablet (Wyeth Pharmaceuticals)

SUMMARY:
The objective of this study was to determine the single-dose bioequivalence of the test product, a potential generic 40 mg pantoprazole delayed-release tablet formulation, compared with the reference product, a pantoprazole 40 mg delayed-release tablet formulation (Protonix, Wyeth Pharmaceuticals), following a single dose in the fasted state.

DETAILED DESCRIPTION:
The 90% CI for pantoprazole ln(Cmax), ln[AUC(0-t)], and ln[AUC(0-inf)] for the comparison of the test product (pantoprazole) versus the reference product (Protonix) should be within the 80 to 125% range required for the conclusion of bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Non tobacco/nicotine-using (6 months minimum) healthy males and females between 19 and 50 years of age.
* Body weight from 15% below or 15% above, inclusive, the ideal weight for height and estimated frame, as adapted from the 1983 Metropolitan Life Table.
* Female subjects were surgically sterile, at least two years postmenopausal, or if sexually active, had a partner who had been vasectomized for at least 6 months, or agreed to utilize one of the following forms of contraception: barrier (condom with spermicide or diaphragm with spermicide), IUD, or hormonal (oral, implant, transdermal patch, or injection) for the following specified times.

Subjects using hormonal contraceptives were on a stable dose for 3 months prior to dosing, or they agreed to also use a barrier method of birth control from screening through completion of the study. Subjects having an intrauterine device (IUD) must have had the IUD in place for at least 2 months prior to dosing, or they agreed to also use a barrier method of birth control from screening through completion of the study. For other forms of birth control, the subject had used the method at least 2 weeks prior to screening and agreed to use the method through completion of the study.

* Voluntary consent to participate in this study as demonstrated by signing the informed consent form.

Exclusion Criteria:

* Persons of Asian origin.
* Females who were pregnant or lactating.
* History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the Investigator, could jeopardize the safety of the subject or impact the validity of the study results.
* History of hypersensitivity, allergic or adverse response to pantoprazole or related drugs.
* Positive results from HIV antibody screen, hepatitis B surface antigen screen, and/or hepatitis C antibody screen.
* Participation in a previous clinical trial within 30 days prior to study initiation.
* Donation of one pint or more of whole blood within 56 days prior to study initiation.
* Donation of 2 units of red blood cells within 112 days prior to study initiation.
* Donation of plasma with 7 days prior to study initiation.
* Difficulty in swallowing medication or any gastrointestinal disease that could affect the drug absorption.
* Abnormal diet or substantial changes in eating habits within 30 days prior to study initiation. Examples included, but were not limited to, vegetarian, fasting, or liquid supplement, etc.
* Treatment with any known enzyme-altering agents (barbiturates, phenothiazines, or cimetidine, etc.) within 30 days prior to study initiation.
* Use of any prescription medication (except hormonal contraceptives for females) within 14 days prior to study initiation.
* Use of any over-the-counter (OTC) medication, including mega-dose vitamins, analgesics, herbal/nutritional supplements, and antacids, within 7 days prior to study initiation.
* Positive urine screen for alcohol or drugs of abuse.
* Unwilling to eat the food as provided in the study menu.
* Hemoglobin <12.0 g/dL.
* History of alcohol or drug abuse within 2 years prior to dosing.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2004-06; Primary Completion 2004-06 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum observed concentration of drug substance in plasma) | 16 hours
AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration) | 16 hours
AUC0-inf area under the concentration-time curve from time zero to infinity) | 16 hoyurs

CONTACTS AND LOCATIONS:
Overall Officials: Alan Marion, MD, PhD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States